CLINICAL TRIAL: NCT03768661
Title: Long-term Incisional Hernia Rate After Single-Incision Laparoscopic Cholecystectomy (SILC) in Front of Standard Laparoscopy
Brief Title: Incisional Hernia Rate After Single-incision Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Hospital Plató (Other)
Responsible Party: Sponsor
Other Study IDs: SILS Chole Hernia
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Cholelithiasis
Keywords: cholecystectomy; laparoscopy; single-incision laparoscopic surgery; incisional hernia; trocar-site hernia
MeSH Terms: conditions — Cholelithiasis; Incisional Hernia | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SILC Group: patients with symptomatic cholelithiasis submitted to a single-incision laparoscopic cholecystectomy
  Interventions: Procedure: Single-incision Laparoscopic cholecystectomy
- Laparoscopy Group: patients with symptomatic cholelithiasis submitted to a standard three trocar laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Single-incision Laparoscopic cholecystectomy — laparoscopic cholecystectomy performed through a single device located at a unique umbilical incision
  Groups: SILC Group
Procedure: Laparoscopic Cholecystectomy — laparoscopic cholecystectomy performed using three-trocars standard technique
  Groups: Laparoscopy Group

SUMMARY:
Single-incision laparoscopic cholecystectomy (SILC) requires a larger incision than standard laparoscopy, which may increase the incidence of incisional hernias.

This study evaluated SILC and standard multiport cholecystectomy with respect to perioperative outcomes, hospital stay, cosmetic results, and postoperative complications, including the 5-years incisional hernia rate.

DETAILED DESCRIPTION:
A cohort study was performed for patients who underwent a laparoscopic cholecystectomy under an institutional review approved protocol. Between 2009 and 2011, 45 unselected patients underwent SILC performed by the same two surgeons.

The study inclusion criteria were the following: patients over 18 years with cholelithiasis, and candidates for elective surgery with no significant cardiopulmonary, hepatic or renal impairment (ASA score less than 4).

The exclusion criteria included the following: acute cholecystitis, associated CBD stones or pancreatitis, an emergency operation for complicated disease, mental illness, or patient refusal and/or absence of informed consent. All included patients signed a standard consent form after being informed about the characteristics of the SILC procedure.

The outcomes of these patients were compared with those of a control cohort series of 140 patients who underwent standard LC (with the same inclusion and exclusion criteria) during the same period.

The primary endpoint of the study was to determine the incisional hernia rate at the umbilical wound after 5 years of follow-up. Hernias were defined as evidence of a hernia at the clinical examination or those confirmed by ultrasound examination in case of clinical doubt.

The study secondary endpoints included the following: duration of surgery (from the start of the incision to skin closure), intraoperative and postoperative complications (30 days), hospital stay, and cosmetic satisfaction results (measured using a visual analogue scale score ranging from 0 to 10).

The following variables were also collected: age, gender, body mass index (BMI) and comorbidities. The anesthetic risk was measured according to the ASA classification system. Prolonged hospital stay (more than 24 h) and readmission (patients who returned for medical consultation before scheduled follow-up) were also recorded. All data were collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years with cholelithiasis and candidates for elective surgery (cholecystectomy)
* abscence of significant cardiopulmonary, hepatic or renal impairment (ASA score less than 4)

Exclusion Criteria:

* acute cholecystitis
* associated common bile duct stones or pancreatitis
* emergency operation for complicated disease
* ASA 4 (American Society of Anesthesiologists)
* pregnancy
* mental illness
* patient refusal and/or absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - patients over 18 years with cholelithiasis and candidates for elective surgery (cholecystectomy)
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
incisional hernia rate | 5 years
  Incisional Hernia by clinical examination or CT scan

SECONDARY OUTCOMES:
operating time of the procedure | During the perioperative period
  Total duration of the surgical procedure (in minutes)
postoperative complications 1 | Rate of participants suffering from biliary complication assesed after 30 days of follow-up
  biliary leak or bile duct injury
postoperative complications 2 | Rate of participants who needed reoperation assesed after 30 days of follow-up
  reoperations
postoperative complications 3 | Rate of participants suffering from seroma and/or wound infection assesed after 30 days of follow-up
  surgical site occurrence
cosmetic satisfaction | patient's own cosmetic evaluation using a visual analogue score ranging from 0 to 10 (0=worst to 10=best) after 30 days of follow-up
  patient's cosmetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hoyuela, MD PhD, Principal Investigator — Chief, Dept. of Surgery
Locations (1):
- Hospital Plató, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoniou SA, Pointner R, Granderath FA. Single-incision laparoscopic cholecystectomy: a systematic review. Surg Endosc. 2011 Feb;25(2):367-77. doi: 10.1007/s00464-010-1217-5. Epub 2010 Jul 7. PMID 20607556
- [Background] Evers L, Bouvy N, Branje D, Peeters A. Single-incision laparoscopic cholecystectomy versus conventional four-port laparoscopic cholecystectomy: a systematic review and meta-analysis. Surg Endosc. 2017 Sep;31(9):3437-3448. doi: 10.1007/s00464-016-5381-0. Epub 2016 Dec 30. PMID 28039641
- [Background] Jorgensen LN, Rosenberg J, Al-Tayar H, Assaadzadeh S, Helgstrand F, Bisgaard T. Randomized clinical trial of single- versus multi-incision laparoscopic cholecystectomy. Br J Surg. 2014 Mar;101(4):347-55. doi: 10.1002/bjs.9393. PMID 24536008
- [Background] Arezzo A, Passera R, Bullano A, Mintz Y, Kedar A, Boni L, Cassinotti E, Rosati R, Fumagalli Romario U, Sorrentino M, Brizzolari M, Di Lorenzo N, Gaspari AL, Andreone D, De Stefani E, Navarra G, Lazzara S, Degiuli M, Shishin K, Khatkov I, Kazakov I, Schrittwieser R, Carus T, Corradi A, Sitzman G, Lacy A, Uranues S, Szold A, Morino M. Multi-port versus single-port cholecystectomy: results of a multi-centre, randomised controlled trial (MUSIC trial). Surg Endosc. 2017 Jul;31(7):2872-2880. doi: 10.1007/s00464-016-5298-7. Epub 2016 Oct 24. PMID 27778171
- [Derived] Hoyuela C, Juvany M, Guillaumes S, Ardid J, Trias M, Bachero I, Martrat A. Long-term incisional hernia rate after single-incision laparoscopic cholecystectomy is significantly higher than that after standard three-port laparoscopy: a cohort study. Hernia. 2019 Dec;23(6):1205-1213. doi: 10.1007/s10029-019-01969-x. Epub 2019 May 9. PMID 31073959
- See also: American Society of Anesthesiologists. ASA Physical Status Classification System — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
- See also: Centers for Disease Control and Prevention. National Healthcare Safety Network (NHSN) Procedure-Associated (PA) Module: Surgical Site Infection (SSI) Event — http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf